CLINICAL TRIAL: NCT03862768
Title: Role of Surgery in Patients With Focally Progressive Gastrointestinal Stromal Tumors (GISTs) After Imatinib Treatment: A Prospective, Multicenter, Randomized Trial
Brief Title: Role of Surgery in Patients With Focally Progressive Gastrointestinal Stromal Tumors (GISTs) After Imatinib Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018-297
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Gastrointestinal Stromal Tumors; Surgery
Keywords: Gastrointestinal Stromal Tumors; imatinib-resistant; focal progression
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Surgical Procedures, Operative; Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery following imatinib (Experimental): Surgery requires at least removal of all drug-resistant lesions. Imatinib 400 MG/d should be taken once the patients resume oral diet.
  Interventions: Procedure: surgery; Drug: Imatinib 400 MG
- Imatinib escalation or sunitinib (Active Comparator): Escalation of imatinib or replacement of sunitinib are both conventional salvage treatments for imatinib-resistant GISTs. There is no high-level evidence to suggest which method is better. So patients are free to choose imatinib 600 MG/d or sunitinib 37.5 MG/d
  Interventions: Drug: Imatinib escalation; Drug: Sunitinib

INTERVENTIONS:
Procedure: surgery — Surgery requires at least removal of all drug-resistant lesions.
  Arms: Surgery following imatinib
Drug: Imatinib 400 MG — Imatinib 400 MG/d should be taken once the patients resume oral diet
  Arms: Surgery following imatinib
Drug: Imatinib escalation — Imatinib 600 MG/d
  Arms: Imatinib escalation or sunitinib
Drug: Sunitinib — Sunitinib 37.5 MG/d
  Arms: Imatinib escalation or sunitinib

SUMMARY:
This study evaluates the efficacy and safety of surgical intervention in patients with focally progressive GISTs after imatinib treatment. The enrolled patients will be randomized to receive surgery following imatinib 400 milligram per day (MG/d) or only tyrosine kinase inhibitor (Imatinib 600 MG/d or Sunitinib 37.5 MG/d).

DETAILED DESCRIPTION:
Imatinib is the first-line treatment for advanced GIST with a satisfactory response rate, but complete remission rarely happens. Besides, drug resistance can occur during the treatment and the median time of drug resistance is about 20-24 months. Once drug resistance occurs, the patient's condition will progress rapidly. As a salvage treatment, the effect of increasing the dose of imatinib or switching to sunitinib is very limited. Progress after imatinib treatment usually involves two conditions, focal progression and extensive progression. For local progression, all resistant lesions can be completely resected; extensive progression refers to resistance progression in multiple sites, and progressive lesions cannot be completely removed. The present study is aimed to assess the benefits of surgical resection of imatinib-resistant lesions in patients with localized disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose pathology is clearly diagnosed as recurrent/metastatic GIST, have undergone standardized imatinib treatment, and the disease progresses during the treatment;
2. The lesions with progress are confined to one organ, and the number is ≤3; after evaluation by relevant professional surgeons or multidisciplinary team discussion, it is considered that the progressive lesions can be completely and safely removed without affecting the organ function;
3. Age: 18 years old ≤ age ≤ 75 years old;
4. No other malignant tumors occurred within five years;
5. Eastern Cooperative Oncology Group (ECOG) physical status score <2 points;
6. American Society of Anesthesiologists (ASA) score <3 points;
7. There are no restrictions on gender and race;
8. Patients with informed consent.

Exclusion Criteria:

1. The patient has other serious comorbidities and cannot tolerate surgery: such as severe cardiopulmonary disease, cardiac function in grade 2 or lower, pulmonary infection, moderate to severe chronic obstructive pulmonary disease (COPD), etc., combined with severe diabetes and/or kidney Insufficient function, combined with severe hepatitis and/or functional Child-pugh grade C or a grade B that is clearly difficult to correct, combined with severe malnutrition;
2. Patients with extensive disease progress;
3. Imatinib primary resistant patients;
4. Patients with other diseases requiring simultaneous surgical intervention, such as gallstones; inguinal hernia;
5. Disease-related complications such as bleeding, perforation, and obstruction;
6. Pregnant or lactating women;
7. The patient has a serious mental illness;
8. Patients with other malignant tumors within five years;
9. The patient has participated in or is participating in other clinical studies or is using other tyrosinekinase inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | one year
  Progression-free survival will be defined as time from the start of treatment until progression (documented according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions) or death, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival | one year
  Overall survival will be defined as time from the start of treatment until death from any cause

IPD SHARING:
Plan to Share IPD: Undecided